CLINICAL TRIAL: NCT03935282
Title: Assessing Effectiveness and Implementation of an EHR Tool to Assess Heart Health Among Survivors (AH-HA)
Brief Title: Assessing Effectiveness and Implementation of an EHR Tool to Assess Heart Health Among Survivors
Acronym: AH-HA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Washington University School of Medicine (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00056774; NCI-2019-01362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA226078 (NIH); NCI-2019-01362 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2019-04-11; First posted 2019-05-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasm; Prostatic Neoplasm; Colorectal Neoplasms; Endometrial Neoplasms; Hodgkin Disease; Non Hodgkin Lymphoma
Keywords: Cardiovascular risk; Cardiovascular disease; Cancer; Survivor; Health Behaviors; Oncology Providers; EHR; Informatics
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Cardiovascular Diseases; Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - AH-HA tool (Experimental): With assistance from the study team, the clinic will implement the AH-HA tool in the clinics' EPIC EHR. Providers at the intervention sites will be trained to use the tool during routine follow-up care with survivors. During a routine follow-up care appointment, the provider will use the AH-HA tool with enrolled patients.
  Interventions: Other: AH-HA Tool in the EPIC EHR
- Usual Care (No Intervention): Usual care practices will conduct routine follow-up care visits for enrolled survivors following typical clinic practice, without use of the AH-HA tool.

INTERVENTIONS:
Other: AH-HA Tool in the EPIC EHR — The Automated Heart-Health Assessment tool implemented in clinics' EPIC EHR will be used by providers during routine follow-up care appointments.
  Arms: Intervention - AH-HA tool

SUMMARY:
The objective of this hybrid effectiveness-implementation study is to examine the effects of an EHR-based cardiovascular health assessment tool (AH-HA) among breast, prostate, colorectal, endometrial, and Hodgkin and non-Hodgkin lymphoma cancer survivors (N=600) receiving survivorship care in community oncology practices, using a group-randomized trial design (6 intervention practices and 6 usual care practices). Our central hypothesis is that the AH-HA tool will increase (1) cardiovascular health (CVH) discussions among survivors and oncology providers, (2) referrals and visits to primary care and cardiology (care coordination), and (3) cardiovascular (CV) risk reduction and health promotion activities compared to usual care.

DETAILED DESCRIPTION:
In this hybrid effectiveness-implementation group-randomized clinical trial, 6 intervention practices will receive an EHR-based cardiovascular health assessment tool (Automated Heart Health Assessment for Survivors: AH-HA) and 6 practices will serve as usual care (control) practices without access to the AH-HA tool. AH-HA renders a visual, interactive display of CVH risk factors, automatically populated from the EHR. This tool was first implemented in primary care and now incorporates EHR data on receipt of cancer treatments with cardiotoxic potential. Providers at each intervention site will be trained to use the tool during routine follow-up care with survivors. Eligible survivors with breast, prostate, colorectal, endometrial, or Hodgkin and non-Hodgkin lymphoma cancer (n=600) will provide baseline data before and immediately after seeing their oncology provider and complete 6-month and 1-year study follow-up visits. The study team will compare changes in outcomes from baseline to 1-year in survivors at the intervention and usual care clinics using data from survivor self-reports and the EHR. The primary outcome is CVH discussions defined as the number of patient-reported discussions with their provider regarding up to seven non-ideal CVH conditions identified for that patient during oncology visits. Secondary outcomes include referrals to primary care and cardiology, provider efforts to manage CV risk, survivors' completed visits with primary care providers and cardiologists, and control of CVH factors and behaviors. Implementation metrics will be assessed using data from the EHR and semi-structured interviews with providers and administrators (n=24-30) at intervention clinics.

ELIGIBILITY:
Inclusion Criteria:

* >= 6 months post-potentially curative cancer treatment for breast, prostate, colorectal, or endometrial cancers or Hodgkin and non-Hodgkin lymphomas. Ongoing hormonal therapies such as tamoxifen, aromatase inhibitors (with or without adjuvant CDK 4/6 inhibitors such as abemaciclib), or androgen deprivation are allowed.
* Scheduled for a routine cancer-related follow-up care visit within the next 30 days with a provider who received training to use AH-HA.
* Able and willing to complete a follow-up assessment in one year.
* Survivors must have no evidence of disease at the time of last medical visit for all cancers, except non-melanoma skin disease.
* Age >= 18 years.
* Able to understand and willing to provide verbal informed consent.

Exclusion Criteria:

* Survivors will be excluded if they have a history of cancer recurrence for any cancer other than non-melanoma skin disease.
* Prostate patients on active surveillance will be excluded.
* Survivor does not speak English or Spanish.
* Survivors who are currently on another interventional protocol in which cardiovascular risk factors (e.g., blood pressure, smoking, diet, physical activity) are being addressed, as per patient self-report or research staff members' knowledge at the time of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least one non-ideal or missing CVH topic | Baseline
  Discussion of non-ideal cardiovascular health (CVH) factors (yes or no). CVH discussions will be defined as patient-reported discussions with their provider for any of the seven non-ideal CVH conditions identified for that patient. Conditions include CVH factors (cholesterol, blood pressure, glucose/hemoglobin A1c) and CVH behaviors (body mass index, smoking, diet, and physical activity). Measured using survivor survey (discussions, diet, and primary care) and EHR for other CVH factors.

SECONDARY OUTCOMES:
Number of referrals to primary care and cardiology to manage CV risk | 1 year
  Medical chart abstraction of referrals and communication with providers regarding CVH at each survivor visit.
Number of CVH-relevant labs and treatments to manage CV risk | 1 year
  Medical chart abstraction.
Completed visits with primary care providers and cardiology | 1 year
  Medical chart abstraction of referrals and communication with providers regarding CVH at each survivor visit.
CVH behaviors recorded in the past year | 1 year
  Medical chart abstraction; Patient survey as secondary, verification source. Measured using smoking status, BMI, physical activity, and healthy diet.
CVH factors recorded in the past year | 1 year
  Medical chart abstraction; Patient survey as secondary, verification source. Measured using total cholesterol, blood pressure, and fasting plasma glucose/Alc.
Patient perception and knowledge of CV risks | Baseline, 6 months, 1 year
  Measured using structured survivor survey. Health knowledge questions were adapted from a survey assessing the relative risk of cancer and cardiovascular disease in United States populations.Minimum score is 0, maximum score is 3 and answer is the total number of questions where a patient responded agree or strongly agree.
Proportion of survivors for whom AH-HA is utilized | 1 year
  We will capture the number of eligible patient visits during which the AH-HA tool was used in intervention clinics and the total number of eligible visits to calculate the proportion of patients where AH-HA was utilized.
Measure of tool acceptability with Tool Assessment | Baseline
  In the Baseline: Post-Visit Survey, survivors will complete a Tool Assessment questionnaire assessing whether or not they recall seeing or discussing the AH-HA tool with their provider and five questions assessing: how much they liked the tool, how helpful it was, how easy it was to understand, how much it improved their understanding, and if they would like to use this tool in the future. Patients will respond to 5 questions on a scale from strongly agree to strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (12):
- United States (12):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration.
Access Criteria: upon request to NCORP@wakehealth.edu

REFERENCES:
- [Background] Shelburne N, Adhikari B, Brell J, Davis M, Desvigne-Nickens P, Freedman A, Minasian L, Force T, Remick SC. Cancer treatment-related cardiotoxicity: current state of knowledge and future research priorities. J Natl Cancer Inst. 2014 Sep 10;106(9):dju232. doi: 10.1093/jnci/dju232. Print 2014 Sep. PMID 25210198
- [Background] Lajous M, Mozaffarian D, Mozaffarian R, Schrag D, Adami HO. Lifestyle prescriptions for cancer survivors and their communities. J Intern Med. 2011 Jan;269(1):88-93. doi: 10.1111/j.1365-2796.2010.02273.x. Epub 2010 Sep 24. PMID 21158981
- [Background] Patnaik JL, Byers T, DiGuiseppi C, Dabelea D, Denberg TD. Cardiovascular disease competes with breast cancer as the leading cause of death for older females diagnosed with breast cancer: a retrospective cohort study. Breast Cancer Res. 2011 Jun 20;13(3):R64. doi: 10.1186/bcr2901. PMID 21689398
- [Background] van Erning FN, van Steenbergen LN, Lemmens VEPP, Rutten HJT, Martijn H, van Spronsen DJ, Janssen-Heijnen MLG. Conditional survival for long-term colorectal cancer survivors in the Netherlands: who do best? Eur J Cancer. 2014 Jul;50(10):1731-1739. doi: 10.1016/j.ejca.2014.04.009. Epub 2014 May 6. PMID 24814358
- [Background] Ward KK, Shah NR, Saenz CC, McHale MT, Alvarez EA, Plaxe SC. Cardiovascular disease is the leading cause of death among endometrial cancer patients. Gynecol Oncol. 2012 Aug;126(2):176-9. doi: 10.1016/j.ygyno.2012.04.013. Epub 2012 Apr 13. PMID 22507532
- [Background] Underwood JM, Townsend JS, Stewart SL, Buchannan N, Ekwueme DU, Hawkins NA, Li J, Peaker B, Pollack LA, Richards TB, Rim SH, Rohan EA, Sabatino SA, Smith JL, Tai E, Townsend GA, White A, Fairley TL; Division of Cancer Prevention and Control, National Center for Chronic Disease Prevention and Health Promotion, Centers for Disease Control and Prevention (CDC). Surveillance of demographic characteristics and health behaviors among adult cancer survivors--Behavioral Risk Factor Surveillance System, United States, 2009. MMWR Surveill Summ. 2012 Jan 20;61(1):1-23. PMID 22258477
- [Background] Foraker RE, Abdel-Rasoul M, Kuller LH, Jackson RD, Van Horn L, Seguin RA, Safford MM, Wallace RB, Kucharska-Newton AM, Robinson JG, Martin LW, Agha G, Hou L, Allen NB, Tindle HA. Cardiovascular Health and Incident Cardiovascular Disease and Cancer: The Women's Health Initiative. Am J Prev Med. 2016 Feb;50(2):236-40. doi: 10.1016/j.amepre.2015.07.039. Epub 2015 Oct 9. PMID 26456876
- [Background] Folsom AR, Yatsuya H, Nettleton JA, Lutsey PL, Cushman M, Rosamond WD; ARIC Study Investigators. Community prevalence of ideal cardiovascular health, by the American Heart Association definition, and relationship with cardiovascular disease incidence. J Am Coll Cardiol. 2011 Apr 19;57(16):1690-6. doi: 10.1016/j.jacc.2010.11.041. PMID 21492767
- [Background] Rasmussen-Torvik LJ, Shay CM, Abramson JG, Friedrich CA, Nettleton JA, Prizment AE, Folsom AR. Ideal cardiovascular health is inversely associated with incident cancer: the Atherosclerosis Risk In Communities study. Circulation. 2013 Mar 26;127(12):1270-5. doi: 10.1161/CIRCULATIONAHA.112.001183. Epub 2013 Mar 18. PMID 23509058
- [Background] Kulshreshtha A, Vaccarino V, Judd SE, Howard VJ, McClellan WM, Muntner P, Hong Y, Safford MM, Goyal A, Cushman M. Life's Simple 7 and risk of incident stroke: the reasons for geographic and racial differences in stroke study. Stroke. 2013 Jul;44(7):1909-14. doi: 10.1161/STROKEAHA.111.000352. Epub 2013 Jun 6. PMID 23743971
- [Background] Hurt RD, Ebbert JO, Hays JT, McFadden DD. Preventing lung cancer by treating tobacco dependence. Clin Chest Med. 2011 Dec;32(4):645-57. doi: 10.1016/j.ccm.2011.08.004. PMID 22054877
- [Background] Byers T, Sedjo RL. Does intentional weight loss reduce cancer risk? Diabetes Obes Metab. 2011 Dec;13(12):1063-72. doi: 10.1111/j.1463-1326.2011.01464.x. PMID 21733057
- [Background] Thomson CA, Rock CL, Thompson PA, Caan BJ, Cussler E, Flatt SW, Pierce JP. Vegetable intake is associated with reduced breast cancer recurrence in tamoxifen users: a secondary analysis from the Women's Healthy Eating and Living Study. Breast Cancer Res Treat. 2011 Jan;125(2):519-27. doi: 10.1007/s10549-010-1014-9. Epub 2010 Jul 6. PMID 20607600
- [Background] Oeffinger KC, Tonorezos ES. The cancer is over, now what?: Understanding risk, changing outcomes. Cancer. 2011 May 15;117(10 Suppl):2250-7. doi: 10.1002/cncr.26051. PMID 21523742
- [Background] Davies NJ, Batehup L, Thomas R. The role of diet and physical activity in breast, colorectal, and prostate cancer survivorship: a review of the literature. Br J Cancer. 2011 Nov 8;105 Suppl 1(Suppl 1):S52-73. doi: 10.1038/bjc.2011.423. PMID 22048034
- [Background] Duprez DA, Otvos J, Sanchez OA, Mackey RH, Tracy R, Jacobs DR Jr. Comparison of the Predictive Value of GlycA and Other Biomarkers of Inflammation for Total Death, Incident Cardiovascular Events, Noncardiovascular and Noncancer Inflammatory-Related Events, and Total Cancer Events. Clin Chem. 2016 Jul;62(7):1020-31. doi: 10.1373/clinchem.2016.255828. Epub 2016 May 12. PMID 27173011
- [Background] Kroenke CH, Chen WY, Rosner B, Holmes MD. Weight, weight gain, and survival after breast cancer diagnosis. J Clin Oncol. 2005 Mar 1;23(7):1370-8. doi: 10.1200/JCO.2005.01.079. Epub 2005 Jan 31. PMID 15684320
- [Background] Caan BJ, Kwan ML, Shu XO, Pierce JP, Patterson RE, Nechuta SJ, Poole EM, Kroenke CH, Weltzien EK, Flatt SW, Quesenberry CP Jr, Holmes MD, Chen WY. Weight change and survival after breast cancer in the after breast cancer pooling project. Cancer Epidemiol Biomarkers Prev. 2012 Aug;21(8):1260-71. doi: 10.1158/1055-9965.EPI-12-0306. Epub 2012 Jun 13. PMID 22695738
- [Background] Jones LW, Haykowsky MJ, Swartz JJ, Douglas PS, Mackey JR. Early breast cancer therapy and cardiovascular injury. J Am Coll Cardiol. 2007 Oct 9;50(15):1435-41. doi: 10.1016/j.jacc.2007.06.037. Epub 2007 Sep 24. PMID 17919562
- [Background] Huffman MD, Capewell S, Ning H, Shay CM, Ford ES, Lloyd-Jones DM. Cardiovascular health behavior and health factor changes (1988-2008) and projections to 2020: results from the National Health and Nutrition Examination Surveys. Circulation. 2012 May 29;125(21):2595-602. doi: 10.1161/CIRCULATIONAHA.111.070722. Epub 2012 Apr 30. PMID 22547667
- [Background] Shay CM, Ning H, Allen NB, Carnethon MR, Chiuve SE, Greenlund KJ, Daviglus ML, Lloyd-Jones DM. Status of cardiovascular health in US adults: prevalence estimates from the National Health and Nutrition Examination Surveys (NHANES) 2003-2008. Circulation. 2012 Jan 3;125(1):45-56. doi: 10.1161/CIRCULATIONAHA.111.035733. Epub 2011 Nov 17. PMID 22095826
- [Background] Byers T, Patnaik JL. Missed opportunities for chronic disease prevention after breast cancer. Womens Health (Lond). 2011 Nov;7(6):619-21. doi: 10.2217/whe.11.66. No abstract available. PMID 22040202
- [Background] Cardinale D, Bacchiani G, Beggiato M, Colombo A, Cipolla CM. Strategies to prevent and treat cardiovascular risk in cancer patients. Semin Oncol. 2013 Apr;40(2):186-98. doi: 10.1053/j.seminoncol.2013.01.008. PMID 23540744
- [Background] Weaver KE, Foraker RE, Alfano CM, Rowland JH, Arora NK, Bellizzi KM, Hamilton AS, Oakley-Girvan I, Keel G, Aziz NM. Cardiovascular risk factors among long-term survivors of breast, prostate, colorectal, and gynecologic cancers: a gap in survivorship care? J Cancer Surviv. 2013 Jun;7(2):253-61. doi: 10.1007/s11764-013-0267-9. Epub 2013 Feb 16. PMID 23417882
- [Background] Christian AH, O'Malley D, Barac A, Miller SM, Hudson SV. Cardiovascular risk and communication among early stage breast cancer survivors. Patient Educ Couns. 2017 Jul;100(7):1360-1366. doi: 10.1016/j.pec.2017.02.010. Epub 2017 Feb 10. PMID 28215826
- [Background] Dennis Parker EA, Sheppard VB, Adams-Campbell L. Compliance with national nutrition recommendations among breast cancer survivors in "stepping stone". Integr Cancer Ther. 2014 Mar;13(2):114-20. doi: 10.1177/1534735413503550. Epub 2013 Oct 7. PMID 24105362
- [Background] Hassoon A, Appel L, Maruthur N and Yeh H-C. Abstract 15582: Cardiovascular Risk Factors in Breast Cancer Survivors: Analysis of NHANES 1999-2012. Circulation. 2015;132:A15582-A15582.
- [Background] Gallicchio L, Calhoun C, Riseberg D, Helzlsouer K. Cardiovascular Health among Black and White Breast Cancer Patients Initiating Aromatase Inhibitor Therapy. Breast J. 2017 Mar;23(2):206-209. doi: 10.1111/tbj.12709. Epub 2016 Oct 25. PMID 27779346
- [Background] Haque R, Prout M, Geiger AM, Kamineni A, Thwin SS, Avila C, Silliman RA, Quinn V, Yood MU. Comorbidities and cardiovascular disease risk in older breast cancer survivors. Am J Manag Care. 2014;20(1):86-92. PMID 24512167
- [Background] Giordano SH, Lin YL, Kuo YF, Hortobagyi GN, Goodwin JS. Decline in the use of anthracyclines for breast cancer. J Clin Oncol. 2012 Jun 20;30(18):2232-9. doi: 10.1200/JCO.2011.40.1273. Epub 2012 May 21. PMID 22614988
- [Background] Bulten BF, Mavinkurve-Groothuis AM, de Geus-Oei LF, de Haan AF, de Korte CL, Bellersen L, van Laarhoven HW, Kapusta L. Early myocardial deformation abnormalities in breast cancer survivors. Breast Cancer Res Treat. 2014 Jul;146(1):127-35. doi: 10.1007/s10549-014-2997-4. Epub 2014 May 23. PMID 24852071
- [Background] Volkova M, Russell R 3rd. Anthracycline cardiotoxicity: prevalence, pathogenesis and treatment. Curr Cardiol Rev. 2011 Nov;7(4):214-20. doi: 10.2174/157340311799960645. PMID 22758622
- [Background] Sawaya H, Sebag IA, Plana JC, Januzzi JL, Ky B, Tan TC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Assessment of echocardiography and biomarkers for the extended prediction of cardiotoxicity in patients treated with anthracyclines, taxanes, and trastuzumab. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):596-603. doi: 10.1161/CIRCIMAGING.112.973321. Epub 2012 Jun 28. PMID 22744937
- [Background] Brana I, Tabernero J. Cardiotoxicity. Ann Oncol. 2010 Oct;21 Suppl 7:vii173-9. doi: 10.1093/annonc/mdq295. PMID 20943611
- [Background] Francis N. The need for routine monitoring of cardiac function in patients receiving 5-fluorouracil infusion. Clin J Oncol Nurs. 2014 Jun;18(3):360-2. doi: 10.1188/14.CJON.360-362. PMID 24867118
- [Background] Meserve EE, Lehmann LE, Perez-Atayde AR, Labelle JL. Cyclophosphamide-associated cardiotoxicity in a child after stem cell transplantation for beta-thalassemia major: case report and review of the literature. Pediatr Dev Pathol. 2014 Jan-Feb;17(1):50-4. doi: 10.2350/13-04-1324-CR.1. Epub 2013 Oct 21. PMID 24144431
- [Background] Khakoo AY, Yeh ET. Therapy insight: Management of cardiovascular disease in patients with cancer and cardiac complications of cancer therapy. Nat Clin Pract Oncol. 2008 Nov;5(11):655-67. doi: 10.1038/ncponc1225. Epub 2008 Sep 16. PMID 18797437
- [Background] Haykowsky MJ, Mackey JR, Thompson RB, Jones LW, Paterson DI. Adjuvant trastuzumab induces ventricular remodeling despite aerobic exercise training. Clin Cancer Res. 2009 Aug 1;15(15):4963-7. doi: 10.1158/1078-0432.CCR-09-0628. Epub 2009 Jul 21. PMID 19622583
- [Background] Saladores P, Murdter T, Eccles D, Chowbay B, Zgheib NK, Winter S, Ganchev B, Eccles B, Gerty S, Tfayli A, Lim JS, Yap YS, Ng RC, Wong NS, Dent R, Habbal MZ, Schaeffeler E, Eichelbaum M, Schroth W, Schwab M, Brauch H. Tamoxifen metabolism predicts drug concentrations and outcome in premenopausal patients with early breast cancer. Pharmacogenomics J. 2015 Feb;15(1):84-94. doi: 10.1038/tpj.2014.34. Epub 2014 Aug 5. PMID 25091503
- [Background] Bird BR, Swain SM. Cardiac toxicity in breast cancer survivors: review of potential cardiac problems. Clin Cancer Res. 2008 Jan 1;14(1):14-24. doi: 10.1158/1078-0432.CCR-07-1033. PMID 18172247
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Darby SC, McGale P, Taylor CW, Peto R. Long-term mortality from heart disease and lung cancer after radiotherapy for early breast cancer: prospective cohort study of about 300,000 women in US SEER cancer registries. Lancet Oncol. 2005 Aug;6(8):557-65. doi: 10.1016/S1470-2045(05)70251-5. PMID 16054566
- [Background] Heidenreich PA, Schnittger I, Strauss HW, Vagelos RH, Lee BK, Mariscal CS, Tate DJ, Horning SJ, Hoppe RT, Hancock SL. Screening for coronary artery disease after mediastinal irradiation for Hodgkin's disease. J Clin Oncol. 2007 Jan 1;25(1):43-9. doi: 10.1200/JCO.2006.07.0805. PMID 17194904
- [Background] Vasu S, Hundley WG. Understanding cardiovascular injury after treatment for cancer: an overview of current uses and future directions of cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jul 31;15(1):66. doi: 10.1186/1532-429X-15-66. PMID 23902649
- [Background] Rock CL, Demark-Wahnefried W. Can lifestyle modification increase survival in women diagnosed with breast cancer? J Nutr. 2002 Nov;132(11 Suppl):3504S-3507S. doi: 10.1093/jn/132.11.3504S. PMID 12421877
- [Background] Singla A, Kumar G, Bardia A. Personalizing cardiovascular disease prevention among breast cancer survivors. Curr Opin Cardiol. 2012 Sep;27(5):515-24. doi: 10.1097/HCO.0b013e3283570040. PMID 22874128
- [Background] Lenihan DJ, Cardinale DM. Late cardiac effects of cancer treatment. J Clin Oncol. 2012 Oct 20;30(30):3657-64. doi: 10.1200/JCO.2012.45.2938. Epub 2012 Sep 24. PMID 23008297
- [Background] Ammon M, Arenja N, Leibundgut G, Buechel RR, Kuster GM, Kaufmann BA, Pfister O. Cardiovascular management of cancer patients with chemotherapy-associated left ventricular systolic dysfunction in real-world clinical practice. J Card Fail. 2013 Sep;19(9):629-34. doi: 10.1016/j.cardfail.2013.07.007. PMID 24054339
- [Background] IOM. Cancer Survivorship Care Planning. 2005.
- [Background] From Cancer Patient to Cancer Survivor: Lost in Transition: The National Academies Press; 2005.
- [Background] Committee on Improving the Quality of Cancer Care: Addressing the Challenges of an Aging Population; Board on Health Care Services; Institute of Medicine; Levit L, Balogh E, Nass S, Ganz PA, editors. Delivering High-Quality Cancer Care: Charting a New Course for a System in Crisis. Washington (DC): National Academies Press (US); 2013 Dec 27. Available from http://www.ncbi.nlm.nih.gov/books/NBK202148/ PMID 24872984
- [Background] Snyder CF, Frick KD, Peairs KS, Kantsiper ME, Herbert RJ, Blackford AL, Wolff AC, Earle CC. Comparing care for breast cancer survivors to non-cancer controls: a five-year longitudinal study. J Gen Intern Med. 2009 Apr;24(4):469-74. doi: 10.1007/s11606-009-0903-2. Epub 2009 Jan 21. PMID 19156470
- [Background] Snyder CF, Earle CC, Herbert RJ, Neville BA, Blackford AL, Frick KD. Trends in follow-up and preventive care for colorectal cancer survivors. J Gen Intern Med. 2008 Mar;23(3):254-9. doi: 10.1007/s11606-007-0497-5. Epub 2008 Jan 16. PMID 18197456
- [Background] Earle CC, Burstein HJ, Winer EP, Weeks JC. Quality of non-breast cancer health maintenance among elderly breast cancer survivors. J Clin Oncol. 2003 Apr 15;21(8):1447-51. doi: 10.1200/JCO.2003.03.060. PMID 12697865
- [Background] Snyder CF, Frick KD, Kantsiper ME, Peairs KS, Herbert RJ, Blackford AL, Wolff AC, Earle CC. Prevention, screening, and surveillance care for breast cancer survivors compared with controls: changes from 1998 to 2002. J Clin Oncol. 2009 Mar 1;27(7):1054-61. doi: 10.1200/JCO.2008.18.0950. Epub 2009 Jan 21. PMID 19164212
- [Background] Weaver KE, Aziz NM, Arora NK, Forsythe LP, Hamilton AS, Oakley-Girvan I, Keel G, Bellizzi KM, Rowland JH. Follow-up care experiences and perceived quality of care among long-term survivors of breast, prostate, colorectal, and gynecologic cancers. J Oncol Pract. 2014 Jul;10(4):e231-9. doi: 10.1200/JOP.2013.001175. Epub 2014 Apr 1. PMID 24695901
- [Background] Emery JD, Shaw K, Williams B, Mazza D, Fallon-Ferguson J, Varlow M, Trevena LJ. The role of primary care in early detection and follow-up of cancer. Nat Rev Clin Oncol. 2014 Jan;11(1):38-48. doi: 10.1038/nrclinonc.2013.212. Epub 2013 Nov 19. PMID 24247164
- [Background] de Moor JS, Mariotto AB, Parry C, Alfano CM, Padgett L, Kent EE, Forsythe L, Scoppa S, Hachey M, Rowland JH. Cancer survivors in the United States: prevalence across the survivorship trajectory and implications for care. Cancer Epidemiol Biomarkers Prev. 2013 Apr;22(4):561-70. doi: 10.1158/1055-9965.EPI-12-1356. Epub 2013 Mar 27. PMID 23535024
- [Background] Daher IN, Daigle TR, Bhatia N, Durand JB. The prevention of cardiovascular disease in cancer survivors. Tex Heart Inst J. 2012;39(2):190-8. PMID 22740730
- [Background] Yang Q, Cogswell ME, Flanders WD, Hong Y, Zhang Z, Loustalot F, Gillespie C, Merritt R, Hu FB. Trends in cardiovascular health metrics and associations with all-cause and CVD mortality among US adults. JAMA. 2012 Mar 28;307(12):1273-83. doi: 10.1001/jama.2012.339. Epub 2012 Mar 16. PMID 22427615
- [Background] Artero EG, Espana-Romero V, Lee DC, Sui X, Church TS, Lavie CJ, Blair SN. Ideal cardiovascular health and mortality: Aerobics Center Longitudinal Study. Mayo Clin Proc. 2012 Oct;87(10):944-52. doi: 10.1016/j.mayocp.2012.07.015. PMID 23036670
- [Background] Xanthakis V, Enserro DM, Murabito JM, Polak JF, Wollert KC, Januzzi JL, Wang TJ, Tofler G, Vasan RS. Ideal cardiovascular health: associations with biomarkers and subclinical disease and impact on incidence of cardiovascular disease in the Framingham Offspring Study. Circulation. 2014 Nov 4;130(19):1676-83. doi: 10.1161/CIRCULATIONAHA.114.009273. Epub 2014 Oct 1. PMID 25274000
- [Background] Cespedes Feliciano EM, Kwan ML, Kushi LH, Weltzien EK, Castillo AL, Caan BJ. Adiposity, post-diagnosis weight change, and risk of cardiovascular events among early-stage breast cancer survivors. Breast Cancer Res Treat. 2017 Apr;162(3):549-557. doi: 10.1007/s10549-017-4133-8. Epub 2017 Feb 7. PMID 28176174
- [Background] Azrad M, Demark-Wahnefried W. The association between adiposity and breast cancer recurrence and survival: A review of the recent literature. Curr Nutr Rep. 2014 Mar;3(1):9-15. doi: 10.1007/s13668-013-0068-9. PMID 24533234
- [Background] Jain R, Strickler HD, Fine E, Sparano JA. Clinical studies examining the impact of obesity on breast cancer risk and prognosis. J Mammary Gland Biol Neoplasia. 2013 Dec;18(3-4):257-66. doi: 10.1007/s10911-013-9307-3. Epub 2013 Nov 13. PMID 24221746
- [Background] Van Blarigan EL, Meyerhardt JA. Role of physical activity and diet after colorectal cancer diagnosis. J Clin Oncol. 2015 Jun 1;33(16):1825-34. doi: 10.1200/JCO.2014.59.7799. Epub 2015 Apr 27. PMID 25918293
- [Background] Fuchs MA, Sato K, Niedzwiecki D, Ye X, Saltz LB, Mayer RJ, Mowat RB, Whittom R, Hantel A, Benson A, Atienza D, Messino M, Kindler H, Venook A, Ogino S, Wu K, Willett WC, Giovannucci EL, Meyerhardt JA. Sugar-sweetened beverage intake and cancer recurrence and survival in CALGB 89803 (Alliance). PLoS One. 2014 Jun 17;9(6):e99816. doi: 10.1371/journal.pone.0099816. eCollection 2014. PMID 24937507
- [Background] Ligibel J. Lifestyle factors in cancer survivorship. J Clin Oncol. 2012 Oct 20;30(30):3697-704. doi: 10.1200/JCO.2012.42.0638. Epub 2012 Sep 24. PMID 23008316
- [Background] Haggstrom DA, Arora NK, Helft P, Clayman ML, Oakley-Girvan I. Follow-up care delivery among colorectal cancer survivors most often seen by primary and subspecialty care physicians. J Gen Intern Med. 2009 Nov;24 Suppl 2(Suppl 2):S472-9. doi: 10.1007/s11606-009-1017-6. PMID 19838853
- [Background] Pearlstein K. Prevalence of cardiovascular disease (CVD) risk factors and preventive care among U.S. cancer survivors. Paper presented at: American Society of Clinical Oncology Annual Meeting; 2013; Chicago, IL.
- [Background] Sharifi M, Adams WG, Winickoff JP, Guo J, Reid M, Boynton-Jarrett R. Enhancing the electronic health record to increase counseling and quit-line referral for parents who smoke. Acad Pediatr. 2014 Sep-Oct;14(5):478-84. doi: 10.1016/j.acap.2014.03.017. PMID 25169159
- [Background] Chrimes D, Kitos NR, Kushniruk A, Mann DM. Usability testing of Avoiding Diabetes Thru Action Plan Targeting (ADAPT) decision support for integrating care-based counseling of pre-diabetes in an electronic health record. Int J Med Inform. 2014 Sep;83(9):636-47. doi: 10.1016/j.ijmedinf.2014.05.002. Epub 2014 May 23. PMID 24981988
- [Background] Zamora A, Fernandez de Bobadilla F, Carrion C, Vazquez G, Paluzie G, Elosua R, Vilaseca M, Martin-Urda A, Rivera A, Plana N, Masana L; VALIDA Study Group; Network of Lipid Units of Catalonia (XULA). Pilot study to validate a computer-based clinical decision support system for dyslipidemia treatment (HTE-DLP). Atherosclerosis. 2013 Dec;231(2):401-4. doi: 10.1016/j.atherosclerosis.2013.09.029. Epub 2013 Oct 18. PMID 24267258
- [Background] Foraker RE, Shoben AB, Kelley MM, Lai AM, Lopetegui MA, Jackson RD, Langan MA, Payne PR. Electronic health record-based assessment of cardiovascular health: The stroke prevention in healthcare delivery environments (SPHERE) study. Prev Med Rep. 2016 Jul 13;4:303-8. doi: 10.1016/j.pmedr.2016.07.006. eCollection 2016 Dec. PMID 27486559
- [Background] Litvin CB, Ornstein SM, Wessell AM, Nemeth LS, Nietert PJ. Use of an electronic health record clinical decision support tool to improve antibiotic prescribing for acute respiratory infections: the ABX-TRIP study. J Gen Intern Med. 2013 Jun;28(6):810-6. doi: 10.1007/s11606-012-2267-2. Epub 2012 Nov 2. PMID 23117955
- [Background] Razavi SA, Carter AB, Puskas JD, Gregg SR, Aziz IF, Buchman TG. Reduced red blood cell transfusion in cardiothoracic surgery after implementation of a novel clinical decision support tool. J Am Coll Surg. 2014 Nov;219(5):1028-36. doi: 10.1016/j.jamcollsurg.2014.06.012. Epub 2014 Jun 25. PMID 25026877
- [Background] Robbins GK, Lester W, Johnson KL, Chang Y, Estey G, Surrao D, Zachary K, Lammert SM, Chueh HC, Meigs JB, Freedberg KA. Efficacy of a clinical decision-support system in an HIV practice: a randomized trial. Ann Intern Med. 2012 Dec 4;157(11):757-66. doi: 10.7326/0003-4819-157-11-201212040-00003. PMID 23208165
- [Background] Kannel WB, D'Agostino RB, Sullivan L, Wilson PW. Concept and usefulness of cardiovascular risk profiles. Am Heart J. 2004 Jul;148(1):16-26. doi: 10.1016/j.ahj.2003.10.022. PMID 15215787
- [Background] Rothman B, Leonard JC, Vigoda MM. Future of electronic health records: implications for decision support. Mt Sinai J Med. 2012 Nov-Dec;79(6):757-68. doi: 10.1002/msj.21351. PMID 23239213
- [Background] Clauser SB, Wagner EH, Aiello Bowles EJ, Tuzzio L, Greene SM. Improving modern cancer care through information technology. Am J Prev Med. 2011 May;40(5 Suppl 2):S198-207. doi: 10.1016/j.amepre.2011.01.014. PMID 21521595
- [Background] Foraker RE, Kite B, Kelley MM, Lai AM, Roth C, Lopetegui MA, Shoben AB, Langan M, Rutledge NL, Payne PR. EHR-based Visualization Tool: Adoption Rates, Satisfaction, and Patient Outcomes. EGEMS (Wash DC). 2015 Jun 18;3(2):1159. doi: 10.13063/2327-9214.1159. eCollection 2015. PMID 26290891
- [Background] Foraker RE, Shoben AB, Lopetegui MA, Lai AM, Payne PR, Kelley M, Roth C, Tindle H, Schreiner A, Jackson RD. Assessment of Life's Simple 7 in the primary care setting: the Stroke Prevention in Healthcare Delivery EnviRonmEnts (SPHERE) study. Contemp Clin Trials. 2014 Jul;38(2):182-9. doi: 10.1016/j.cct.2014.03.007. Epub 2014 Apr 8. PMID 24721482
- [Background] HIMSS. United States EMR Adoption Model. EMR Adoption Model. 2012.
- [Background] Mamlin BW, Tierney WM. The Promise of Information and Communication Technology in Healthcare: Extracting Value From the Chaos. Am J Med Sci. 2016 Jan;351(1):59-68. doi: 10.1016/j.amjms.2015.10.015. PMID 26802759
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Alzaman N, Wartak SA, Friderici J, Rothberg MB. Effect of patients' awareness of CVD risk factors on health-related behaviors. South Med J. 2013 Nov;106(11):606-9. doi: 10.1097/SMJ.0000000000000013. PMID 24192590
- [Background] McDonald M, Hertz RP, Unger AN, Lustik MB. Prevalence, awareness, and management of hypertension, dyslipidemia, and diabetes among United States adults aged 65 and older. J Gerontol A Biol Sci Med Sci. 2009 Feb;64(2):256-63. doi: 10.1093/gerona/gln016. Epub 2009 Jan 30. PMID 19181717
- [Background] Miles A, Simon A, Wardle J. Answering patient questions about the role lifestyle factors play in cancer onset and recurrence: what do health care professionals say? J Health Psychol. 2010 Mar;15(2):291-8. doi: 10.1177/1359105309351245. PMID 20207672
- [Background] Jones LW, Courneya KS, Fairey AS, Mackey JR. Effects of an oncologist's recommendation to exercise on self-reported exercise behavior in newly diagnosed breast cancer survivors: a single-blind, randomized controlled trial. Ann Behav Med. 2004 Oct;28(2):105-13. doi: 10.1207/s15324796abm2802_5. PMID 15454357
- [Background] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948
- [Background] Reeves MM, Terranova CO, Eakin EG, Demark-Wahnefried W. Weight loss intervention trials in women with breast cancer: a systematic review. Obes Rev. 2014 Sep;15(9):749-68. doi: 10.1111/obr.12190. Epub 2014 May 29. PMID 24891269
- [Background] Winters-Stone KM, Beer TM. Review of exercise studies in prostate cancer survivors receiving androgen deprivation therapy calls for an aggressive research agenda to generate high-quality evidence and guidance for exercise as standard of care. J Clin Oncol. 2014 Aug 10;32(23):2518-9. doi: 10.1200/JCO.2014.55.8189. Epub 2014 Jul 7. No abstract available. PMID 25002711
- [Background] Hawkes AL, Chambers SK, Pakenham KI, Patrao TA, Baade PD, Lynch BM, Aitken JF, Meng X, Courneya KS. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. J Clin Oncol. 2013 Jun 20;31(18):2313-21. doi: 10.1200/JCO.2012.45.5873. Epub 2013 May 20. PMID 23690410
- [Background] Zbikowski SM, Magnusson B, Pockey JR, Tindle HA, Weaver KE. A review of smoking cessation interventions for smokers aged 50 and older. Maturitas. 2012 Feb;71(2):131-41. doi: 10.1016/j.maturitas.2011.11.019. Epub 2011 Dec 29. PMID 22209349
- [Background] Stead LF, Bergson G, Lancaster T. Physician advice for smoking cessation. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000165. doi: 10.1002/14651858.CD000165.pub3. PMID 18425860
- [Background] Improving Cancer-Related Outcomes with Connected Health: A Report to the President of the United States from the President's Cancer Panel. 2016.
- [Background] Chang VW, Lauderdale DS. Fundamental cause theory, technological innovation, and health disparities: the case of cholesterol in the era of statins. J Health Soc Behav. 2009 Sep;50(3):245-60. doi: 10.1177/002214650905000301. PMID 19711804
- [Background] Highland KB, Hurtado-de-Mendoza A, Stanton CA, Dash C, Sheppard VB. Risk-reduction opportunities in breast cancer survivors: capitalizing on teachable moments. Support Care Cancer. 2015 Apr;23(4):933-41. doi: 10.1007/s00520-014-2441-7. Epub 2014 Sep 21. PMID 25239599
- [Background] Bluethmann SM, Mariotto AB, Rowland JH. Anticipating the "Silver Tsunami": Prevalence Trajectories and Comorbidity Burden among Older Cancer Survivors in the United States. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1029-36. doi: 10.1158/1055-9965.EPI-16-0133. PMID 27371756
- [Background] Howlader N, Noone A, Krapcho M, Garshell J, Miller D, Altekruse S, Kosary C, Yu M, Ruhl J, Tatalovich Z, Mariotto A, Lewis D, Chen H, Feuer E and Cronin K. SEER Cancer Statistics Review, 1975-2011. SEER. 2014.
- [Background] Kessler RS, Purcell EP, Glasgow RE, Klesges LM, Benkeser RM, Peek CJ. What does it mean to "employ" the RE-AIM model? Eval Health Prof. 2013 Mar;36(1):44-66. doi: 10.1177/0163278712446066. Epub 2012 May 21. PMID 22615498
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] RE-AIM. Reach Effectiveness Adoption Implementation Maintenance. 2017;2017.
- [Background] Arora NK, Reeve BB, Hays RD, Clauser SB, Oakley-Girvan I. Assessment of quality of cancer-related follow-up care from the cancer survivor's perspective. J Clin Oncol. 2011 Apr 1;29(10):1280-9. doi: 10.1200/JCO.2010.32.1554. Epub 2011 Feb 28. PMID 21357781
- [Background] Lloyd-Jones DM, Hong Y, Labarthe D, Mozaffarian D, Appel LJ, Van Horn L, Greenlund K, Daniels S, Nichol G, Tomaselli GF, Arnett DK, Fonarow GC, Ho PM, Lauer MS, Masoudi FA, Robertson RM, Roger V, Schwamm LH, Sorlie P, Yancy CW, Rosamond WD; American Heart Association Strategic Planning Task Force and Statistics Committee. Defining and setting national goals for cardiovascular health promotion and disease reduction: the American Heart Association's strategic Impact Goal through 2020 and beyond. Circulation. 2010 Feb 2;121(4):586-613. doi: 10.1161/CIRCULATIONAHA.109.192703. Epub 2010 Jan 20. PMID 20089546
- [Background] Centers for Medicare & Medicaid Services (CMS), HHS. HIPAA administrative simplification: National Plan and Provider Enumeration System Data Dissemination. Notice. Fed Regist. 2007 May 30;72(103):30011-4. PMID 17577966
- [Background] Murray DM, Pals SL, Blitstein JL, Alfano CM, Lehman J. Design and analysis of group-randomized trials in cancer: a review of current practices. J Natl Cancer Inst. 2008 Apr 2;100(7):483-91. doi: 10.1093/jnci/djn066. Epub 2008 Mar 25. PMID 18364501
- [Background] Murray DM, Varnell SP, Blitstein JL. Design and analysis of group-randomized trials: a review of recent methodological developments. Am J Public Health. 2004 Mar;94(3):423-32. doi: 10.2105/ajph.94.3.423. PMID 14998806
- [Background] Eldridge SM, Ashby D, Feder GS, Rudnicka AR, Ukoumunne OC. Lessons for cluster randomized trials in the twenty-first century: a systematic review of trials in primary care. Clin Trials. 2004 Feb;1(1):80-90. doi: 10.1191/1740774504cn006rr. PMID 16281464
- [Background] Smith JJ, Morgan PJ, Plotnikoff RC, Dally KA, Salmon J, Okely AD, Finn TL, Babic MJ, Skinner G, Lubans DR. Rationale and study protocol for the 'active teen leaders avoiding screen-time' (ATLAS) group randomized controlled trial: an obesity prevention intervention for adolescent boys from schools in low-income communities. Contemp Clin Trials. 2014 Jan;37(1):106-19. doi: 10.1016/j.cct.2013.11.008. Epub 2013 Nov 26. PMID 24291151
- [Background] Sandelowski M, Leeman J. Writing usable qualitative health research findings. Qual Health Res. 2012 Oct;22(10):1404-13. doi: 10.1177/1049732312450368. Epub 2012 Jun 28. PMID 22745362
- [Background] Foraker R, Kelley M, Wilkister T, Lin E-J and Weaver K. Oncologists' perceptions of the usability of SPHERE: an electronic health record applicaton based on Life's Simple 7. American Heart Association. 2016;133:AP075.
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Background] Mosca L, Jones WK, King KB, Ouyang P, Redberg RF, Hill MN. Awareness, perception, and knowledge of heart disease risk and prevention among women in the United States. American Heart Association Women's Heart Disease and Stroke Campaign Task Force. Arch Fam Med. 2000 Jun;9(6):506-15. doi: 10.1001/archfami.9.6.506. PMID 10862212
- [Derived] Nightingale CL, Dressler EV, Kepper M, Klepin HD, Lee SC, Smith S, Aguilar A, Wiseman KD, Sohl SJ, Wells BJ, DeMari JA, Throckmorton A, Kulbacki LW, Hanna J, Foraker RE, Weaver KE. Oncology Provider and Patient Perspectives on a Cardiovascular Health Assessment Tool Used During Posttreatment Survivorship Care in Community Oncology (Results from WF-1804CD): Mixed Methods Observational Study. J Med Internet Res. 2025 Mar 6;27:e65152. doi: 10.2196/65152. PMID 39854647
- [Derived] Weaver KE, Dressler EV, Klepin HD, Lee SC, Wells BJ, Smith S, Hundley WG, Lesser GJ, Nightingale CL, Turner JC, Lackey I, Heard K, Foraker R; AH-HA Study Team. Effectiveness of a Cardiovascular Health Electronic Health Record Application for Cancer Survivors in Community Oncology Practice: Results From WF-1804CD. J Clin Oncol. 2025 Jan;43(1):46-56. doi: 10.1200/JCO.24.00342. Epub 2024 Nov 21. PMID 39571113
- [Derived] Weaver KE, Dressler EV, Smith S, Nightingale CL, Klepin HD, Lee SC, Wells BJ, Hundley WG, DeMari JA, Price SN, Foraker RE. Cardiovascular health assessment in routine cancer follow-up in community settings: survivor risk awareness and perspectives. BMC Cancer. 2024 Jan 31;24(1):158. doi: 10.1186/s12885-024-11912-8. PMID 38297229
- [Derived] DeMari JA, Dressler EV, Foraker RE, Wells BJ, Smith S, Klepin H, Hundley WG, Lesser GJ, Shalowitz DI, Nightingale CL, Hernandez M, Weaver KE. Endometrial cancer survivors' perceptions of their cardiovascular disease risk (results from WF-1804CD AH-HA). Gynecol Oncol. 2023 Jul;174:208-212. doi: 10.1016/j.ygyno.2023.05.009. Epub 2023 May 22. PMID 37224793

DOCUMENTS (1):
  • Informed Consent Form (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03935282/ICF_000.pdf